CLINICAL TRIAL: NCT04726982
Title: Optimal Dosage of Acetazolamide for Obstructive Sleep Apnea Treatment: a Parallel-group, Double-blind, Placebo-controlled, Randomized Trial
Brief Title: Optimal Dosage of Acetazolamide for OSA Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B3002021000015
Record Dates: First submitted 2021-01-26; First posted 2021-01-27 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: Carbonic anhydrase inhibitor; Treatment; Pharmacotherapy; Sleep apnea; Loop gain; Respiration; Ventilatory control instability; Acidosis
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Respiratory Aspiration; Acidosis | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose acetazolamide (Experimental): Unembellished white tablets. The drug should be taken one hour before bedtime. Total treatment duration will be 6 weeks.
  Interventions: Drug: Acetazolamide
- High dose acetazolamide (Experimental): Unembellished white tablets. The drug should be taken one hour before bedtime. Total treatment duration will be 6 weeks.
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Matching placebo tablets. The drug should be taken one hour before bedtime. Total treatment duration will be 6 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acetazolamide — 250 mg once daily
  Other Names: Diamox; ATC code: S01EC01
  Arms: Low dose acetazolamide
Drug: Acetazolamide — 500 mg once daily
  Other Names: Diamox; ATC code: S01EC01
  Arms: High dose acetazolamide
Other: Placebo — Once daily
  Arms: Placebo

SUMMARY:
Acetazolamide, a carbonic anhydrase inhibitor, has received some attention as potential treatment for obstructive sleep apnea (OSA). It produces a metabolic acidosis by excreting bicarbonate, thereby stimulating baseline ventilation. Evidence suggests that acetazolamide primarily improves ventilatory control instability (expressed as loop gain), which is an important contributor to the pathophysiology of OSA.

Few studies have assessed the efficacy of acetazolamide in patients with OSA. Since most of them had a small sample size and used different therapeutic dosages, clinical applications are currently limited. Therefore, this study aims to compare the effect of two acetazolamide dosages on the severity and pathophysiology of OSA.

DETAILED DESCRIPTION:
In this double-blind, parallel-group, controlled trial, eligible patients will be randomized into one of the following treatment arms: (1) placebo, (2) 250 mg of acetazolamide, or (3) 500 mg of acetazolamide. After 4 weeks, treatment outcome will be assessed by in-laboratory polysomnography. Additionally, arterial blood gas analysis and lung function tests will be performed before and during treatment.

ELIGIBILITY:
Inclusion Criteria:

* AHI between 15 and 65 events/hour
* BMI < 35 kg/m²

Exclusion Criteria:

* Craniofacial anomalies
* Central sleep apnea (defined as central AHI > 25% of total AHI)
* Contra-indications related to acetazolamide treatment

  * Hypersensitivity to sulphonamides or acetazolamide
  * Renal impairment, electrolyte imbalances, and/or adrenocortical insufficiency
  * Clinically significant metabolic, hepatic, and/or hematological disease
  * Chronic obstructive pulmonary disease
  * Closed-angle glaucoma
* Conditions likely to affect OSA physiology: neuromuscular disease or other major neurological disorders, heart failure, or any other unstable major medical condition.
* Intake of drugs that substantially stimulate or depress respiration, including benzodiazepines, opioids, theophylline, and pseudoephedrine
* Inadequately treated sleep disorders other than OSA that would confound functional sleep assessment
* Inability of the patient to understand and/or comply to the study procedures
* Active psychiatric disease (psychotic illness, major depression, anxiety attacks, alcohol or drug abuse)
* Pregnancy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | 4 weeks
  Change in AHI (events/hour) from baseline to follow-up. The AHI is a measure of sleep apnea severity that encompasses the frequency of apneas (cessations in breathing) and hypopneas (reductions in airflow).

SECONDARY OUTCOMES:
Pathophysiological traits | 4 weeks
  Changes in pathophysiological traits (Vpassive, Vactive, Arousal Threshold, Loop Gain) will be quantified as %Veupnea from polysomnography data using a validated algorithm.
Percent responders | 4 weeks
  Treatment response will be defined as a reduction in AHI of ≥ 50%.
Nocturnal oxygen saturation | 4 weeks
  Change in mean and minimal SaO2 (%).
Oxygen desaturation index (ODI) | 4 weeks
  Change in ODI (events/hour) from baseline to follow-up. The ODI represents the average number of desaturation episodes (≥ 3%) per hour sleep.
Arterial blood gas measurements | 4 weeks
  Change in pO2 (mmhg) and pCO2 (mmhg) from baseline to follow-up.
Lung function parameters | 4 weeks
  Change in flow-volume curve from baseline to follow-up.
Daytime sleepiness: Epworth Sleepiness Scale (ESS) | 6 weeks
  The ESS asks respondents to rate on a 4-point scale (0-3) their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores) can range from 0 to 24. The higher the ESS score, the higher that person's sleep propensity in daily life. A score higher than 10 indicates the presence of excessive daytime sleepiness.
Sleep-related quality of life: Functional Outcome of Sleep Questionnaire (FOSQ-10) | 6 weeks
  This questionnaire is an abbreviated version of the original 30-item version. The FOSQ-10 consists of 10 items that are distributed among 5 subscales: general productivity (2 items), activity level (3 items), vigilance (3 items), social outcomes (1 item), and intimacy and sexual relationships (1 item). The questionnaire has a 4-point scale. The total score is calculated as the sum of the subscale means and can range from 5 to 20. The minimal important difference ranges from 1.7 to 2.0 points.
Snoring intensity: Visual Analogue Scale (VAS) | 6 weeks
  A standard 10-point VAS ranging from 0 (no snoring) to 10 (extreme snoring) will be used to evaluate the subjective status of snoring during sleep. Heavy snoring corresponds to a snoring index of at least 7. A decrease of 3 points after treatment is considered significant. To be considered as an important reduction, snoring needs to reduce to an index that is no longer experienced as bothersome (i.e. < 3).

OTHER OUTCOMES:
Incidence of adverse events | 6 weeks
  Safety and tolerability of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Vanderveken, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No